CLINICAL TRIAL: NCT07108179
Title: Continuous Glucose Monitoring System: Accuracy and Prognostic Value in Critically Ill Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Sinocare (Industry)
Responsible Party: Sponsor
Other Study IDs: SN-CGM-PO-002
Record Dates: First submitted 2025-07-25; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-01

CONDITIONS: Critically Ill Patients
MeSH Terms: interventions — Continuous Glucose Monitoring; Drug Delivery Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Continuous Glucose Monitoring (CGM) System — Continuous Glucose Monitoring (CGM) System

SUMMARY:
Whether diabetic or non-diabetic patients, blood glucose management during ICU hospitalization is essential. This study aims to evaluate the accuracy of the iCan Continuous Glucose Monitoring (CGM) System for detecting blood glucose levels in ICU patients, as well as its value in prognostic evaluation, to provide reference for blood glucose management in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years; gender not limited.
2. Expected ICU (Intensive Care Unit) stay ≥ 48 hours.
3. Patients requiring frequent blood gas monitoring in the ICU.

Exclusion Criteria:

1. The patient or their family refuses to use CGM for blood glucose monitoring.
2. Patients with adverse skin conditions (such as rash, active inflammation, etc.) in the device placement area, or those requiring emergency surgical intervention in that area.
3. Patients who need to undergo computed tomography (CT), X-ray, or magnetic resonance imaging (MRI) scans on the device placement area during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Accuracy | Up to eight days
  "Comparison between arterial blood gas analysis glucose values and CGM values at the same time"

CONTACTS AND LOCATIONS:
Locations (1):
- Continuous glucose monitoring system, Changsha, changsha, China

IPD SHARING:
Plan to Share IPD: No